CLINICAL TRIAL: NCT05272761
Title: Impact of Breathing Route on the Effectiveness of Treatment of Obstructive Sleep Apnea With CPAP and Oronasal Mask
Brief Title: Impact of Breathing Route on CPAP Effectiveness to Treat Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, Principal Investigator, University of Sao Paulo General Hospital
Other Study IDs: 4901/19/120
Record Dates: First submitted 2021-12-28; First posted 2022-03-09 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: OSA; Apnea+Hypopnea
Keywords: Breathing route; OSA; CPAP; Oronasal mask; Apnea hypopnea index; Air leak; Sleep efficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oronasal Route: Patients will sleep in the sleep lab for CPAP titration wearing a custom oronasal mask with 2 open oral and nasal compartments. The titration was split between the first half of the night and the second half. The titration will be started with the patient remaining for 90 minutes with the pressure he uses at home (supine position and in lateral decubitus), after a period of 90 minutes the patient will be titrated in order to abolish respiratory events in both positions of the body.
- Oral Route: Group/Cohort Interventions Oronasal Route
  Patients will sleep in the sleep lab for CPAP titration using a custom 2-compartment oronasal mask. In this titration, the nasal compartment will be closed and the patient will be titrated only through the oral route. The titration split between the first half of the night and the second half. The titration will be started with the patient staying for 90 minutes with the pressure used at home (during the supine position and lateral position), after the 90 minute period the patient will be titrated in order to abolish respiratory events in both positions of the body.

SUMMARY:
To determine the impact of the CPAP route (oronasal vs oral) in patients diagnosed with moderate-severe OSA using CPAP with oronasal mask on CPAP level, residual AHI, and peak flow. In addition, the impact of position (lateral vs supine position) will be evaluated during PSG.

DETAILED DESCRIPTION:
Application of Continuous Positive Upper Airway Pressure (CPAP) during sleep using nasal mask is the gold standard treatment for Obstructive Sleep Apnea (OSA). In clinical practice, many patients with OSA are considered mouth breathers and use an oronasal mask. However, CPAP delivered by the mouth violates the principal of CPAP use to treat OSA. This study is part of a line of research over the last decade that started with the observation of a patient that CPAP delivered by an oronasal mask failed to splint the airway open and to abolish OSA . We showed subsequently in acute studies during induced-sleep that oronasal CPAP only works when the patient breathes predominantly through the nose. These observations prompted our group to lead one workshop on the importance of mask selection. One meta-analysis from our group confirmed that oronasal CPAP is associated with a higher CPAP level, higher residual AHI, and poorer adherence than nasal CPAP. Despite all this evidence the investigators intrigued by the clinical observation that oronasal masks remains common and several patients on clinical practice are well adapted to oronasal CPAP. In this study, 20 patients with OSA well adapted to the oronasal mask will be recruited. The patients will be invited to be submitted to 2 independent CPAP titration sleep studies using a customized oronasal mask with a sealed and independent nasal and oral compartments coupled to 2 pneumotachographs. One CPAP titration will be with the nasal and oral routes open and one CPAP titration with only the oral compartment opened. Our hypotheses are that obstruction of nasal compartment during CPAP titration causuing mouth breathing will result in higher CPAP and higher residual apnea-hypopnea index. Patients with OSA under treatment with oronasal CPAP will undergo CPAP titration polysomnography on 2 different nights. In one night the patient will sleep with the oral and nasal compartments opened and in another night interposed by at least seven days, the patient with sleep with only the oral compartment opened. The order of the 2 sleep studies will be randomized. Thus, researchers will assess the impact of the airway (oral vs oronasal) on titrated CPAP level, residual AHI, and sleep efficiency in supine and lateral recumbency. In addition, the preferred airway during the oronasal mask will be analyzed. At the end of the study a nasal mask will be offered to all patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate or severe OSA in treatment with CPAP in an oronasal mask
* 18 Years to 85 Years (Adult, Older Adult) (Adult, Older Adult)

Exclusion Criteria:

* Other sleep disturbance (insomnia, parasomnias, narcolepsy, central sleep apnea).
* Uncontrolled clinical disease (diabetes, kidney or heart failure, recent stroke or coronary failure and recent postoperative period, oxygen dependent COPD).
* Patients adapted to other types of masks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis moderate or severe OSA in treatment with CPAP in an Oronasal Mask
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-02-18 (Estimated)

PRIMARY OUTCOMES:
Impact of breathing route on residual AHI | 2 nights
  To determine the impact of the CPAP route (oronasal vs oral) in patients diagnosed with moderate-severe OSA using oronasal mask on residual AHI ( Apnea-hypopnea Index).
Impact of breathing route on the CPAP | 2 nights
  To determine the impact of the CPAP route (oronasal vs oral) in patients during titration of the CPAP route (oronasal vs oral)

SECONDARY OUTCOMES:
Influence of position | 2 nights
  To assess the influence of body position on the CPAP pressure used at home by the patient in the oral and oronasal route.

CONTACTS AND LOCATIONS:
Overall Officials: Geraldo Lorenzi-Filho, PHD, Principal Investigator — Hospital das Clínicas HCFMUSP
Locations (1):
- Fundação Zerbini - Instituto do Coração (InCor), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Schorr F, Genta PR, Gregorio MG, Danzi-Soares NJ, Lorenzi-Filho G. Continuous positive airway pressure delivered by oronasal mask may not be effective for obstructive sleep apnoea. Eur Respir J. 2012 Aug;40(2):503-5. doi: 10.1183/09031936.00145111. No abstract available. PMID 22855472
- [Background] Andrade RG, Madeiro F, Piccin VS, Moriya HT, Schorr F, Sardinha PS, Gregorio MG, Genta PR, Lorenzi-Filho G. Impact of Acute Changes in CPAP Flow Route in Sleep Apnea Treatment. Chest. 2016 Dec;150(6):1194-1201. doi: 10.1016/j.chest.2016.04.017. Epub 2016 Apr 29. PMID 27132703
- [Background] Madeiro F, Andrade RGS, Piccin VS, Pinheiro GDL, Moriya HT, Genta PR, Lorenzi-Filho G. Transmission of Oral Pressure Compromises Oronasal CPAP Efficacy in the Treatment of OSA. Chest. 2019 Dec;156(6):1187-1194. doi: 10.1016/j.chest.2019.05.024. Epub 2019 Jun 22. PMID 31238041
- [Background] Genta PR, Kaminska M, Edwards BA, Ebben MR, Krieger AC, Tamisier R, Ye L, Weaver TE, Vanderveken OM, Lorenzi-Filho G, DeYoung P, Hevener W, Strollo P. The Importance of Mask Selection on Continuous Positive Airway Pressure Outcomes for Obstructive Sleep Apnea. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2020 Oct;17(10):1177-1185. doi: 10.1513/AnnalsATS.202007-864ST. PMID 33000960
- [Background] Andrade RGS, Viana FM, Nascimento JA, Drager LF, Moffa A, Brunoni AR, Genta PR, Lorenzi-Filho G. Nasal vs Oronasal CPAP for OSA Treatment: A Meta-Analysis. Chest. 2018 Mar;153(3):665-674. doi: 10.1016/j.chest.2017.10.044. Epub 2017 Dec 19. PMID 29273515
- [Derived] Xavier JLA, Fernandes MD, Andrade RGS, Genta PR, Lorenzi-Filho G. Impact of Exclusive Mouth Route and Lateral Position on the Efficacy of Oronasal CPAP to Treat OSA in Patients With OSA Adapted to Oronasal Mask. Chest. 2025 Feb;167(2):611-618. doi: 10.1016/j.chest.2024.10.023. Epub 2024 Oct 24. PMID 39454998